CLINICAL TRIAL: NCT00381017
Title: A Randomized, Open-label, Multi-center, Phase 3, 2-arm Study Evaluating the Efficacy and Safety of Peg Interferon Alfa-2b Low-dose Maintenance Monotherapy Versus Standard Supportive Care in Patients With Cirrhotic Hepatitis C Co-infected With Human Immunodeficiency Virus - The ENDURE Study
Brief Title: Effects of Low-dose Maintenance Peg Interferon Alfa-2b Therapy Versus Supportive Care in Patients With Cirrhotic Hepatitis C With HIV (Study P04371)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Non-protocol feasibility
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Integrated Therapeutics Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04371; EUDRACT NUMBER:2005-003876-39
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Hepatitis C; Liver Cirrhosis; HIV Infections
MeSH Terms: conditions — Hepatitis C; Liver Cirrhosis; HIV Infections | interventions — peginterferon alfa-2b

INTERVENTIONS:
Drug: Peg interferon alpha-2b

SUMMARY:
This is a Phase 3b, randomized, open-label, parallel-group, multi-center, multi-national study of low-dose maintenance Peg interferon alpha-2b (Peg-Intron®) in subjects with human immunodeficiency virus-hepatitis C virus (HIV-HCV) co-infection. The primary objective is to compare at end of study the efficacy of Peg-Intron® monotherapy (0.5 µg/kg subcutaneously once weekly for 24-36 months) versus standard supportive care, using the time to any of the following clinical events (death, decompensation, liver transplant, hepatocellular carcinoma [HCC]) as endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years but < 70 years, of either sex or any race.
* Detectable plasma hepatitis C virus (HCV) RNA (all genotypes of HCV are permitted).
* Cirrhosis of the liver within the last five years.
* Compensated liver disease (Child-Pugh <8 with hepatic encephalopathy <= 1.
* No evidence of hepatocellular carcinoma (HCC) and a serum alpha fetoprotein (AFP) <100 ng/mL within two months of randomization/study enrollment.
* Varices results via endoscopy within the last six months or at time of screening.
* Serologic evidence of human immunodeficiency virus-1.
* CD4 cell count >=100 /µL.
* Platelet number of at least 50000 mm**3.
* Neutrophil count of at least 750 mm**3.
* Hemoglobin of >9.0 mg%.
* Serum thyroid stimulating hormone levels within normal limits, regardless of treatment with L thyroxin.
* Hemoglobin A1c (HbA1c)<8.5%, to demonstrate controlled diabetes, if applicable.
* Written clearance from an ophthalmologist must be presented for subjects with a history of hypertension or diabetes prior to treatment start.
* Creatinine clearance >50 mL/min, as assessed by the indirect calculation method.
* Demonstrate stable status of HIV-1 infection.
* On stable antiretroviral therapy (HAART) for at least 6 weeks prior to baseline, with the expectation of their HAART regimen (drugs and dosage) remaining unaltered for the first 8 weeks of the study OR
* Willing to delay initiation of HAART therapy for at least 6 weeks (for subjects who have not been on HAART for at least 8 weeks prior to randomization). "Structured treatment interruptions" will be permitted during the study.
* Counseled in the appropriate use of birth control while in this study, as confirmed by the principal investigator or a sub-investigator.
* Free of any clinically significant disease (other than HCV and HIV) that would interfere with study evaluations.

Exclusion Criteria:

* Female who is pregnant, intends to become pregnant during the study or within two months after study completion, or is nursing. Male subject whose partner wants to become pregnant.
* Using silymarin.
* Positive test at screening for anti-HAV IgM Ab, HBsAg, anti-HBc IgM Ab, or HBeAg.
* Any cause of liver disease other than chronic hepatitis C.
* Suspected or having hypersensitivity to interferon.
* History of liver decompensation status or other evidence of bleeding from esophageal varices, signs of current bleeding, significant ascites, hepatic encephalopathy, jaundice or other conditions consistent with decompensated liver disease.
* Present with a lesion suspicious for hepatic malignancy on the screening imaging.
* Any active malignant disease, suspicion, or history of malignant disease within 5 years prior to study enrollment (except for adequately treated basal cell carcinoma).
* Known coagulation or hemoglobin diseases.
* Organ transplant, except corneal or hair transplant.
* Any known preexisting medical condition that, in the investigator's opinion, could interfere with the subject's participation in and completion of the study, such as major depressive disorder.
* Active HIV-related opportunistic infection and/or malignancy requiring systemic therapy.
* Evidence of known severe retinopathy.
* Subject has not observed the designated washout periods for any of the prohibited medications.
* Participating in any other hepatitis C clinical study.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-09